CLINICAL TRIAL: NCT02636673
Title: Robotic-assisted Versus Laparoscopic Sigmoid Resection: a Retrospective Chart Review of Benign and Malignant Sigmoid Disease
Brief Title: Robotic-assisted Versus Laparoscopic Sigmoid Resection
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVSR-001
Record Dates: First submitted 2015-12-07; First posted 2015-12-22 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Sigmoid Diseases
MeSH Terms: conditions — Sigmoid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robotic-assisted sigmoid resection: Patient that have undergone robotic-assisted sigmoid resection for benign or malignant disease between 2010 and 2015
  Interventions: Procedure: Sigmoid Resection
- Laparoscopic sigmoid resection: Patient that have undergone laparoscopic sigmoid resection for benign or malignant disease between 2010 and 2015
  Interventions: Procedure: Sigmoid Resection

INTERVENTIONS:
Procedure: Sigmoid Resection

SUMMARY:
Retrospective multi-center comparative chart review of robotic-assisted versus laparoscopic sigmoid resection for both benign and malignant disease

DETAILED DESCRIPTION:
The goal is to establish safety and effectiveness of robotic-assisted surgery in sigmoid resection for both benign and malignant disease by evaluation of short-term clinical outcomes through 30 days post index procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients that have undergone sigmoid resection for benign or malignant disease

Exclusion Criteria:

* Emergency Procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects that have undergone robotic-assisted or laparoscopic sigmoid resection for benign and malignant disease will be considered for inclusion except those that had emergency procedures.
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of complications observed intraoperatively through 30-days | Intraoperative through 30-days follow-up
  Number of complications observed intraoperatively through 30-days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - HonorHealth / Colon & Rectal Clinic of Scottsdale, Scottsdale, Arizona
  - Jackson South Community Hospital, Miami, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Progressive Surgical Associates/Silver Cross Hospital, New Lenox, Illinois
  - Northern Weschester Hospital, Mount Kisco, New York
  - Aria Health, Phildelphia, Pennsylvania